CLINICAL TRIAL: NCT06171646
Title: Effect of Breathing Exercise on Fatigue in Patients With Pulmonary Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sema Aytaç, PhD (Network)
Responsible Party: Sponsor-Investigator, Sema Aytaç, PhD, Asist Prof. Dr, Tuberculosis Network European Trialsgroup
Organization: Tuberculosis Network European Trialsgroup (Network)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5122023
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis, Pulmonary; Fatigue
MeSH Terms: conditions — Tuberculosis, Pulmonary; Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental, Breathing Group (Experimental): Breathing exercises were applied to the participants.
  Interventions: Behavioral: breathing exercise
- No Intervention: Standard care (No Intervention): Participants received standard care.

INTERVENTIONS:
Behavioral: breathing exercise — The patients in the intervention group will first be informed by the researcher about pursed lips and diaphragmatic breathing exercises through a face-to-face interview technique, and then the breathing exercises will be taught practically to each patient for approximately 30 minutes, and the first session will be held. Each session takes place once a day in the morning, lasts 10-15 minutes and is applied every day; Sessions other than the first session will consist of 10 pursed lip breathing exercises, relaxation (2 minutes) and 10 diaphragmatic breathing exercises; Three days a week, the researcher will be reminded via online video call once a day in the morning, and on the other days, the patients will be reminded by phone call that they will be asked to do themselves, and breathing exercises will be performed for a total of four weeks.
  Arms: Experimental, Breathing Group

SUMMARY:
Tuberculosis is a chronic, necrotic infectious disease with very different clinical appearances, caused by a group of mycobacteria defined as M. tuberculosis complex. Although there is a vaccine and can be treated with combined medications, this health problem remains important all over the world, especially in poor countries. Generally, respiratory symptoms that occur in a person with tuberculosis include cough, phlegm, hemoptysis, chest pain, and shortness of breath for more than three weeks. If there is a partial obstruction in the bronchi due to the compression of enlarged lymph nodes, it causes a whezing sound accompanied by shortness of breath. In tuberculosis, contagion is brought under control with effective treatment by regular use of drugs. In addition, the symptoms of the patients are relieved until they recover. However, the fatigue of the patients may continue. The disease may continue. In addition to having an effect, fatigue may also occur due to the side effects of many tuberculosis drugs. Therefore, patients experiencing fatigue while taking tuberculosis drugs may cause them to become uncooperative in drug use, multidrug-resistant tuberculosis, serious complications and higher treatment costs. Another method used in addition to the treatment of chronic respiratory system diseases such as tuberculosis is pulmonary rehabilitation.Pulmonary rehabilitation consists of patient education, psychosocial support, aerobic and strengthening breathing exercises and physical training programs. Among the breathing exercises that are considered to be one of the important components of pulmonary rehabilitation, pursed-lip breathing and diaphragmatic breathing exercises are frequently used in chronic respiratory system diseases. However, no study has been found examining the effects of pursed-lip breathing and diaphragmatic breathing exercises on fatigue in tuberculosis patients. Pursed-lip breathing technique ensures maximum emptying of the alveoli by providing controlled expiration, thus helping to reduce the respiratory rate by increasing the activity of the inspiratory and expiratory muscles, increasing gas exchange and tidal volume. During diaphragmatic breathing exercise, since the diaphragm muscle is used instead of accessory muscles, the respiratory load decreases, thus the ventilation level of the lungs increases and breathing is supported. It has been reported in the literature that the deep breathing technique is effective in controlling the emotional states of tuberculosis patients, and that deep breathing exercises applied to pulmonary TB patients are effective in reducing the respiratory rate. However, since no study was found in the literature review that evaluated the effect of breathing exercise applied to TB patients on fatigue, this study was planned to examine the effect of breathing exercise applied to patients diagnosed with TB on fatigue.

ELIGIBILITY:
Inclusion Criteria:

Being literate Being diagnosed with Pulmonary Tuberculosis and completing the 15th day of treatment Volunteering to participate in the study Being 18 years or older No communication problems Not having mental confusion or any psychiatric problems Not having Multiple Drug Resistance (MDR) Using a communication tool

Exclusion Criteria:

Reluctance to participate in the study Being a patient with Multiple Drug Resistance (MDR) Not being diagnosed with Pulmonary Tuberculosis and not having completed the 15th day of treatment Having any psychiatric problems Scoring '0' on the Piper Fatigue scale Not using communication tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in fatigue during the Follow-up | 1 months
  Piper fatigue scale was applied. It varies between 0-10 points, with a higher score indicating increased fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No